CLINICAL TRIAL: NCT03797248
Title: The Clinical Outcome of Adjuvant Chemotherapy in Conjunction With Traditional Chinese Medicine in Breast Cancer Patients -a Observational Cohort Study
Brief Title: Prospective Cohort Study of Traditional Chinese Medicine for Survival of Patients With Early Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ming-Yen Tsai, Department of Chinese medicine, Chang Gung Memorial Hospital
Other Study IDs: 201801559A3
Record Dates: First submitted 2019-01-05; First posted 2019-01-09 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Early-stage Breast Cancer
Keywords: traditional Chinese medicine; quality of life; disease-free survival; adjuvant chemotherapy; breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: adjuvant chemotherapy combined with Chinese herbal medicine
  Interventions: Combination Product: Chinese herbal medicine
- Cohort 2: adjuvant chemotherapy only
  Interventions: Combination Product: Chinese herbal medicine

INTERVENTIONS:
Combination Product: Chinese herbal medicine — All Chinese herbal products prescribed from TCM physicians in our hospital during patients receiving adjuvant chemotherapy

SUMMARY:
This 2-year trial is intended to be used to study breast cancer patients through forward-looking generation design through collaboration between Chinese and Western medical teams. The whole study consists of 2 stages, stage I comprises a cross-sectional study-baseline and stage II is a cohort for outcome evaluation and follow-up study across a 3-year period. To provide an empirical basis for combined TCM treatment in the Breast Cancer Research Team and to publish that as a reference for future TCM and Western medicine in integrative cancer treatment.

DETAILED DESCRIPTION:
Breast cancer is a major health issue for women worldwide and has increased exponentially in the last decades. Improved earlier detection combined with adjuvant systemic therapy is responsible for much of the reduction in cause-specific mortality from breast cancer. Chemotherapy after surgery can decrease the risk of recurrence and is often used as routine treatment in clinic. Because of the fact that a considerable number of patients seek for traditional Chinese medicine (TCM) during adjuvant chemotherapy, it is thus need to evaluate the correlation between TCM treatment and prognosis. The investigators design a single center, prospective cohort study began in November 2018 in Kaohsiung, Taiwan. A sample of 104 participants diagnosed with early breast cancer was recruited from Breast Cancer Research Team and are followed up every 3 to 6 months till October 2023. Detailed information of participants includes general information, history of cancer, quality of life, side effects of chemotherapy and safety of treatment, body constitution of TCM and meridian energy analysis is taken face-to-face at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Aged > 20 years old female patients;
* Patients with histologically proven stage 1-3 breast cancer after surgery;
* The duration from the end of radical surgery to the beginning of the trail is less than 1 month;
* ECOG score is 0-2 points;
* Agreed to participate in this study and signed informed consent.

Exclusion Criteria:

* Combined with inadequate heart, liver, kidney and hematopoietic function and other serious diseases;
* Pregnant and lactating women;
* Patients with a history of mental illness;
* Patients with distant metastasis and/or expected lifetime less than 3 months;
* Patients undergoing other medicinal herbs outside our hospital.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with breast cancer aged over 20 years with histologically diagnosed stage 1-3 after radical surgery are enrolled from an academic medical center. All participants need to complete the 6-8 cycle of adjuvant chemotherapy, which may last 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 310 (Estimated)
Dates: Start 2018-11-12 (Actual); Primary Completion 2020-10-24 (Estimated); Study Completion 2020-10-24 (Estimated)

PRIMARY OUTCOMES:
disease-free survival | 3 years
  3-year disease-free survival

SECONDARY OUTCOMES:
QOLs measurement-1 | 6 months
  Functional Assessment of Cancer Therapy - Breast Cancer(FACT-B)
QOLs measurement-2 | 6 months
  Eastern Cooperative Oncology Group (ECOG)
TCM pattern | 6 months
  Body Constitution Questionnaire (BCQ)
meridian energy | 6 months
  Meridian Energy Analysis Device (MEAD)
Side effects of adjuvant chemotherapy | 6 months
  Common Terminology Criteria for Adverse Events (CTCAE)

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Ting Liu, MD, Principal Investigator — Division of Oncology, Department of Internal Medicine
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No
The datasets during and/or analyzed during the current study available from the corresponding author on reasonable request.

REFERENCES:
- [Derived] Liu CT, Chen YH, Huang YC, Chen SY, Tsai MY. Chemotherapy in conjunction with traditional Chinese medicine for survival of patients with early female breast cancer: protocol for a non-randomized, single center prospective cohort study. Trials. 2019 Dec 17;20(1):741. doi: 10.1186/s13063-019-3848-8. PMID 31847861